CLINICAL TRIAL: NCT03974880
Title: Predicting the Clinical Outcomes of Patients With Lower Extremity Peripheral Arterial Disease Undergoing Endovascular Intervention Based on Computed Tomographic Angiography
Brief Title: Predicting Outcomes of PAD Patients Undergoing Endovascular Intervention With CTA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2019LSY-16
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patency group: Freedom from restenosis or clinically driven re-intervention in the treated lesion at 1,3,6,12 months after procedures
- restenosis group: Restenosis was defined as a reduction in the luminal diameter of more than 50 percent according to any imaging examinations such as duplex ultrasound, CTA, MRI or DSA Re-intervention in the treated segment for the clinical progression at 1,3,6,12 months after procedures
- the second adverse events group: a composite of all-cause death, myocardial infarction, and stroke and any amputation at 1,3,6,12 months after procedures

SUMMARY:
Lower extremity peripheral artery disease (PAD), the third leading cause of atherosclerotic cardiovascular morbidity following coronary artery disease and stroke, affect 200 million people worldwide and is associated with high rates of cardiovascular events and death. Consensus is reached on an "endovascular-first-strategy" for symptomatic PAD who have developed critical limb ischemia.

However, the challenge of endovascular therapy is the long-term patency, and the associated worse clinical outcomes, including higher rates of major adverse cardiovascular events, and major adverse limb events. Meta-analysis concluded that restenosis occurred rate 5-70 % at 1 year; the incidence of adverse limb outcomes, (including worsening of symptoms, the need for peripheral revascularization, and amputation) was 26% over a period of 4 years; Cardiovascular morbidity and mortality up to 28 % after endovascular therapy.

There are no consensus guidelines on the optimal timing and the factor on adverse clinical outcome remains uncertain. Therefore, the purpose of this study is to conduct a structured surveillance plan for follow-up care and evaluate risk factors that will eventually support development of a predictive model for clinical outcomes of endovascular procedures to treat lower extremity PAD.

DETAILED DESCRIPTION:
This is a prospective, observational, multi-center, clinical study examining predictors of clinical outcomes for patients undergoing PAD endovascular treatment. The study population will undergo lower extremity computed tomographic angiography (CTA )and endovascular intervention procedures. CT scanning was performed with the coverage from the common iliac artery bifurcation to the tiptoe, CTA data were transfer to an offline workstation for further analysis. Axial images, cross-sectional views, curved planar reformations and multiplane reformations, as well as three dimensional maximum intensity projection images were available for evaluation. This includes disease in a vessel located proximal(involving the aortoiliac and femoropopliteal locations), distal, (involving the infrapopliteal location), proximal and distal (multilevel disease).

We conduct a detailed chart review to gather the data related to the index endovascular intervention procedures report, study personnel history and physical presentation, laboratory inspection, the lesion characteristics arising from CTA. Data abstract from chart review include indication for procedure (intermittent claudication, rest pain, and tissue loss), detailed lesion characteristics (lesion length, stenosis severity, diameter, and presence of total occlusion), procedure(s) performed and devices used, and per procedural events.

Patients will be followed up for the occurrence of these outcomes from the time of their initial revascularization procedure(1month after enrollment, and at months 3 (+- 2 weeks), 6 (+- 2 weeks), and 12 (+- 2 weeks)).

The follow-up of Clinical outcomes : Primary clinical outcomes of interest were ：1）restenosis in the treated segment（Restenosis was defined as a reduction in the luminal diameter of more than 50 percent according to any imaging examinations such as duplex ultrasound, CTA,magnetic resonance Imaging(MRI) or digital subtraction angiography(DSA) ）；2）re-intervention in the treated segment for the clinical progression. Secondary end points included:1) all lower extremity amputation, 2) all -cause death, myocardial infarction, and stroke; 3) a neo- segment more than 75 % stenosis and clinical assessment requires intervention .

Cox proportional hazards models were created to show the hazard ratios (HRs) associated with lesion characters and patient demographic and clinical characteristics ,and further identify predictors of clinical outcomes, moreover, plotted unadjusted Kaplan Meier curves for lower extremity peripheral artery patients undergone endovascular revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age ≥ 18 years.
2. Subject presents with a Fontaine classification of 2 to 5;
3. Subject presents with clinical evidence of PAD requiring endovascular intervention on one or both limbs that includes a target lesion, and never undergo endovascular intervention on any limb.

If subject presents with bilateral disease, the first limb treated with a lesion in the target area will be considered the target limb.

Exclusion Criteria:

1. Subject is unwilling or unable to sign the informed consent form.
2. Subject is unable to understand or comply with the study protocol requirements.
3. Subject has been performed a surgical bypass graft for any lesion(s) in the target area or amputation as determined by the Investigator.
4. Subject has a history of malignant tumor.
5. The interval between CTA and endovascular intervention is more than 1 month and the CTA images could not be evaluated because of motion and metal artifact.
6. Subject has the contraindications to CTA or DSA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAD patients met the inclusion criteria underwent pre-procedue CTA and endovascular revascularization
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
restenosis group | at 1,3,6,12 moth
  Restenosis was defined as a reduction in the luminal diameter of more than 50 percent according to any imaging examinations such as duplex ultrasound, CTA, MRI or DSA
re-intervention group | at 1,3,6,12 moth
  re-intervention in the treated segment for the clinical progression, but a reduction in the luminal diameter of low than 50 percent according to any imaging examinations.

SECONDARY OUTCOMES:
amputation | at 1,3,6,12 moth
  all lower extremity amputation
Co-morbid cardio-cerebral vascular diseases | at 1,3,6,12 moth
  Co-morbid cardio-cerebral vascular diseases include all -cause death, myocardial infarction, and stroke
neo- segment lesion | at 1,3,6,12 moth
  a neo- segment lesion is more than 75 % stenosis and clinical assessment requires intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yang, MD,PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes